CLINICAL TRIAL: NCT00309790
Title: Phase 3 Study of the Effects of Chronic Sildenafil Citrate Therapy on Exercise Tolerance and Hemodynamics in Patients With Advanced Heart Failure.
Brief Title: Study of Sildenafil in Advanced Heart Failure.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Marc J Semigran, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-p-0003994
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Congestive Heart Failure
Keywords: exercise stress test
MeSH Terms: conditions — Heart Failure | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil

SUMMARY:
Despite advances in medical therapy for patients with heart failure, one-third of patients remain limited by fatigue and shortness of breath.

Our previous study concluded that one dose of sildenafil (Viagra) lead to an improvement in heart pressure and exercise capacity.

Currently sildenafil is not FDA approved for the treatment of heart failure.

The purpose of this study is to determine if treatment with sildenafil for 12 weeks in patients with heart failure can improve exercise capacity and quality of life in people with heart failure.

DETAILED DESCRIPTION:
This study will compare two groups of patients. One group will receive sildenafil and the other group will receive a placebo (a pill which looks like sildenafil, but contains no medication).

Patients will undergo a heart catheterization, echocardiogram and exercise stress test. Patients will then take study medication for 12 weeks. A repeat heart catheterization, echocardiogram and exercise stress test will then be performed.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years Ejection fraction <40% Heart failure limited by fatigue and shortness of breath Pulmonary artery hypertension

Exclusion Criteria:

Patients taking the following medications: nitroglycerine pill/patch/paste, isordil, Imdur, antifungal agents and certain antidepressants.

Patients with a history of optic neuropathy or unexplained visual impairment. Patients with anemia.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-05; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Patients will have the following performed at baseline and again after taking study medication for 12 weeks: exercise capacity measured by exercise stress test, heart pressure measured by a heart catheterization and
quality of life measured by questionnaires at baseline and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Semigran, MD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Derived] Malhotra R, Dhakal BP, Eisman AS, Pappagianopoulos PP, Dress A, Weiner RB, Baggish AL, Semigran MJ, Lewis GD. Pulmonary Vascular Distensibility Predicts Pulmonary Hypertension Severity, Exercise Capacity, and Survival in Heart Failure. Circ Heart Fail. 2016 Jun;9(6):10.1161/CIRCHEARTFAILURE.115.003011 e003011. doi: 10.1161/CIRCHEARTFAILURE.115.003011. PMID 27301469
- [Derived] Murphy RM, Shah RV, Malhotra R, Pappagianopoulos PP, Hough SS, Systrom DM, Semigran MJ, Lewis GD. Exercise oscillatory ventilation in systolic heart failure: an indicator of impaired hemodynamic response to exercise. Circulation. 2011 Sep 27;124(13):1442-51. doi: 10.1161/CIRCULATIONAHA.111.024141. Epub 2011 Aug 29. PMID 21875912
- [Derived] Lewis GD, Murphy RM, Shah RV, Pappagianopoulos PP, Malhotra R, Bloch KD, Systrom DM, Semigran MJ. Pulmonary vascular response patterns during exercise in left ventricular systolic dysfunction predict exercise capacity and outcomes. Circ Heart Fail. 2011 May;4(3):276-85. doi: 10.1161/CIRCHEARTFAILURE.110.959437. Epub 2011 Feb 3. PMID 21292991